CLINICAL TRIAL: NCT04636814
Title: A 52-week, Randomized, Double-blind, Double-dummy, Placebo- and Active- Controlled (Roflumilast, Daliresp® 500µg), Parallel Group, Study to Evaluate the Efficacy and Safety of Two Doses of CHF6001 DPI add-on to Maintenance Triple Therapy in Subjects With Chronic Obstructive Pulmonary Disease (COPD) and Chronic Bronchitis.
Brief Title: A 52-week, Placebo- and Active- Controlled (Roflumilast, Daliresp® 500µg) Study to Evaluate the Efficacy and Safety of Two Doses of CHF6001 DPI (Tanimilast) as add-on to Maintenance Triple Therapy in Subjects With COPD and Chronic Bronchitis. (PILLAR)
Acronym: PILLAR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic decision by Sponsor; not due to safety reasons
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLI-06001AA1-05; 2020-003648-97 (EudraCT Number); 2023-510174-13-00 (EU CTIS Number)
Record Dates: First submitted 2020-11-16; First posted 2020-11-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; chronic bronchitis; PDE4 inhibitor; anti-inflammatory respiratory drug; Tanimilast
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — tanimilast; Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CHF6001 1600µg (Experimental)
  Interventions: Drug: CHF6001 1600µg
- CHF6001 3200µg (Experimental)
  Interventions: Drug: CHF6001 3200µg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Roflumilast (Active Comparator)
  Interventions: Drug: Roflumilast

INTERVENTIONS:
Drug: CHF6001 1600µg — CHF6001 400µg, 2 inhalations bid (total daily dose of 1600µg) and Roflumilast matching placebo, 1 tablet once daily
  Arms: CHF6001 1600µg
Drug: CHF6001 3200µg — CHF6001 800µg, 2 inhalations bid (total daily dose of 3200µg) and Roflumilast matching placebo, 1 tablet once daily
  Arms: CHF6001 3200µg
Drug: Placebo — CHF6001 matching placebo, 2 inhalations bid and Roflumilast matching placebo, 1 tablet once daily
  Arms: Placebo
Drug: Roflumilast — - 1 tablet of Roflumilast (Daliresp®), 250µg, once daily during the first 4 weeks of treatment then 1 tablet of Roflumilast (Daliresp®), 500µg, once daily for the remaining treatment period and CHF6001 matching placebo, 2 inhalations bid
  Arms: Roflumilast

SUMMARY:
The purpose of this study is to evaluate the efficacy and the safety of two doses of CHF6001 (Tanimilast) as add-on to maintenance triple therapy in the target patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 40 years, with COPD and with chronic bronchitis.
* Current smokers or ex-smokers (history of ≥10 pack years).
* Post-bronchodilator FEV1 <50% of the patient predicted normal value and FEV1/FVC ratio < 0.7.
* At least, one moderate or severe COPD exacerbation in the previous year.
* CAT score ≥10.
* Subjects on regular maintenance triple therapy for at least 12 months prior to screening and receiving regular maintenance triple therapy for at least 3 months prior to screening visit.

Exclusion Criteria:

* Subjects with current asthma.
* Subjects with moderate or severe COPD exacerbation 4 weeks before study entry and randomisation
* Subjects with known α-1 antitrypsin deficiency as the underlying cause of COPD.
* Subjects with primary diagnosis of emphysema not related to COPD.
* Subjects with known respiratory disorders other than COPD.
* Subjects with lung volume reduction surgery.
* Subjects with active cancer or a history of lung cancer.
* Subjects under Roflumilast treatment within 6 months before study entry.
* Subjects with a diagnosis of depression, generalised anxiety disorder, suicidal ideation.
* Subjects with clinically significant cardiovascular condition.
* Subjects with neurological disease.
* Subjects with clinically significant laboratory abnormalities.
* Subjects with moderate or severe hepatic impairment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3973 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
The number of moderate and severe exacerbations occurring during the planned 52-week treatment period. | Up to 52 weeks
  Moderate or severe exacerbation is defined by symptomatic worsening of COPD:
  * Moderate : requiring use of systemic corticosteroids (oral/IV/IM corticosteroids), and/or use of antibiotics
  * Severe : requiring hospitalisation or resulting in death

SECONDARY OUTCOMES:
The time to first moderate or severe exacerbation. | Up to 52 weeks
  The time to first moderate or severe exacerbation.
The annual rate of severe exacerbations. | Up to 52 weeks
  The annual rate of severe exacerbations.
The time to first severe exacerbation. | Up to 52 weeks
  The time to first severe exacerbation.
The number of all on-treatment severe exacerbations. | Up to 52 weeks
  The number of all on-treatment severe exacerbations.
The number of all on-treatment exacerbations requiring systemic corticosteroids. | Up to 52 weeks
  The number of all on-treatment exacerbations requiring systemic corticosteroids.
Change from baseline (pre-dose Visit 2) in pre-dose FEV1, at week 52. | At week 52
  Change from baseline (pre-dose Visit 2) in pre-dose FEV1, at week 52.
Change from baseline in Saint Georges Respiratory Questionnaire (SGRQ) total and domain scores at week 52. | At week 52
  Change from baseline in Saint Georges Respiratory Questionnaire (SGRQ) total and domain scores at week 52.
Saint Georges Respiratory Questionnaire response (SGRQ) (change from baseline SGRQ total score ≤ -4) at week 52. | At week 52
  Saint Georges Respiratory Questionnaire response (SGRQ) (change from baseline SGRQ total score ≤ -4) at week 52.
Change from baseline to last inter-visit period (week 40-52) in EXACT-Respiratory Symptoms (E-RS) Total and subscale scores. | Up to 52 weeks
  Change from baseline to last inter-visit period (week 40-52) in EXACT-Respiratory Symptoms (E-RS) Total and subscale scores.
E-RS response (change from baseline E-RS Total score ≤ -2) at week 52. | At week 52
  E-RS response (change from baseline E-RS Total score ≤ -2) at week 52.
Change from baseline to last inter-visit period (week 40-52) in the percentage of days without intake of rescue medication and in the average rescue medication use (number of puffs). | Up to 52 weeks
  Change from baseline to last inter-visit period (week 40-52) in the percentage of days
Time to study medication discontinuation for any reason. | Up to 52 weeks
  Time to study medication discontinuation for any reason.
Time to moderate or severe exacerbation or study medication discontinuation due to any adverse event, lack of efficacy or death (composite endpoint) and time to study medication discontinuation component. | Up to 52 weeks
  Time to moderate or severe exacerbation or study medication discontinuation due to any adverse event, lack of efficacy or death (composite endpoint) and time to study medication discontinuation component.
Time to first moderate/severe exacerbation or study medication discontinuation due to any class-related AE, lack of efficacy, or death (composite endpoint) and time to study medication discontinuation component. | Up to 52 weeks
  Time to first moderate/severe exacerbation or study medication discontinuation due to any class-related AE, lack of efficacy, or death (composite endpoint) and time to study medication discontinuation component.
Key Secondary Variable: Change from baseline in SGRQ Total score at week 52 | At week 52
  Key Secondary Variable: Change from baseline in SGRQ Total score at week 52

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J. MARTINEZ, Prof., Principal Investigator — Weill Cornell Medical College, New York Presbyterian Hospital, 1305 York avenue box 96 NY 10021 USA
Locations (460):
- United States (150):
  - Chiesi Clinical Trial - Site 840635, Andalusia, Alabama
  - Chiesi Clinical Trial - Site 840614, Foley, Alabama
  - Chiesi Clinical Trial - Site 840670, Guntersville, Alabama
  - Chiesi Clinical Trial - Site 840720, Mobile, Alabama
  - Chiesi Clinical Trial - Site 840643, Saraland, Alabama
  - Chiesi Clinical Trial - Site 840638, Phoenix, Arizona
  - Chiesi Clinical Trial - Site 840684, Conway, Arkansas
  - Chiesi Clinical Trial - Site 840675, Laguna Hills, California
  - Chiesi Clinical Trial - Site 840666, Los Angeles, California
  - Chiesi Clinical Trial - Site 840511, Newport Beach, California
  - Chiesi Clinical Trial - Site 840680, Northridge, California
  - Chiesi Clinical Trial - Site 840605, Northridge, California
  - Chiesi Clinical Trial - Site 840700, Pomona, California
  - Chiesi Clinical Trial - Site 840531, Westminster, California
  - Chiesi Clinical Trial - Site 840636, Centennial, Colorado
  - Chiesi Clinical Trial - Site 840688, Lakewood, Colorado
  - Chiesi Clinical Trial - Site 840735, Brooksville, Florida
  - Chiesi Clinical Trial - Site 840513, Chiefland, Florida
  - Chiesi Clinical Trial - Site 840652, Clearwater, Florida
  - Chiesi Clinical Trial - Site 840569, Clearwater, Florida
  - Chiesi Clinical Trial - Site 840545, Coral Gables, Florida
  - Chiesi Clinical Trial - Site 840603, Cutler Bay, Florida
  - Chiesi Clinical Trial - Site 840587, Cutler Bay, Florida
  - Chiesi Clinical Trial - Site 840568, Cutler Bay, Florida
  - Chiesi Clinical Trial - Site840539, Daytona Beach, Florida
  - Chiesi Clinical Trial - Site 840554, DeBary, Florida
  - Chiesi Clinical Trial - Site 840625, Doral, Florida
  - Chiesi Clinical Trial - Site 840572, Doral, Florida
  - Chiesi Clinical Trial - Site 840685, Hialeah, Florida
  - Chiesi Clinical Trial - Site 840504, Hialeah, Florida
  - Chiesi Clinical Trial - Site 840639, Hialeah, Florida
  - Chiesi Clinical Trial - Site 840582, Hialeah, Florida
  - Chiesi Clinical Trial - Site 840617, Hialeah, Florida
  - Chiesi Clinical Trial - Site 840514, Hialeah, Florida
  - Chiesi Clinical Trial - Site 840637, Hialeah Gardens, Florida
  - Chiesi Clinical Trial - Site 840509, Hollywood, Florida
  - Chiesi Clinical Trial - Site 840730, Hollywood, Florida
  - Chiesi Clinical Trial - Site 840565, Homestead, Florida
  - Chiesi Clinical Trial - Site 840674, Loxahatchee Groves, Florida
  - Chiesi Clinical Trial - Site 840732, Melbourne, Florida
  - Chiesi Clinical Trial - Site 840624, Miami, Florida
  - Chiesi Clinical Trial - Site 840596, Miami, Florida
  - Chiesi Clinical Trial - Site 840556, Miami, Florida
  - Chiesi Clinical Trial - Site 840602, Miami, Florida
  - Chiesi Clinical Trial - Site 840507, Miami, Florida
  - Chiesi Clinical Trial - Site 840519, Miami, Florida
  - Chiesi Clinical Trial - Site 840505, Miami, Florida
  - Chiesi Clinical Trial - Site 840644, Miami, Florida
  - Chiesi Clinical Trial - Site 840557, Miami, Florida
  - Chiesi Clinical Trial - Site 840588, Miami, Florida
  - Chiesi Clinical Trial - Site 840618, Miami, Florida
  - Chiesi Clinical Trial - Site 840525, Miami, Florida
  - Chiesi Clinical Trial - Site 840656, Miami, Florida
  - Chiesi Clinical Trial - Site 840622, Miami, Florida
  - Chiesi Clinical Trial - Site 840537, Miami, Florida
  - Chiesi Clinical Trial - Site 840691, Miami, Florida
  - Chiesi Clinical Trial - Site 840503, Miami, Florida
  - Chiesi Clinical Trial - Site 840694, Miami, Florida
  - Chiesi Clinical Trial - Site 840630, Miami, Florida
  - Chiesi Clinical Trial - Site 840506, Miami Gardens, Florida
  - Chiesi Clinical Trial - Site 840608, Miami Lakes, Florida
  - Chiesi Clinical Trial - Site 840524, Orlando, Florida
  - Chiesi Clinical Trial - Site 840563, Orlando, Florida
  - Chiesi Clinical Trial - Site 840702, Pembroke Pines, Florida
  - Chiesi Clinical Trial - Site 840502, Pembroke Pines, Florida
  - Chiesi Clinical Trial - Site 840550, Pembroke Pines, Florida
  - Chiesi Clinical Trial - Site 840527, Pompano Beach, Florida
  - Chiesi Clinical Trial - Site 840654, South Miami, Florida
  - Chiesi Clinical Trial - Site 840699, St. Petersburg, Florida
  - Chiesi Clinical Trial - Site 840697, St. Petersburg, Florida
  - Chiesi Clinical Trial - Site 840567, Tampa, Florida
  - Chiesi Clinical Trial - Site 840632, Winter Park, Florida
  - Chiesi Clinical Trial - Site 840542, Adairsville, Georgia
  - Chiesi Clinical Trial - Site 840728, College Park, Georgia
  - Chiesi Clinical Trial - Site 840717, Columbus, Georgia
  - Chiesi Clinical Trial - Site 840710, Cordele, Georgia
  - Chiesi Clinical Trial - Site 840689, East Point, Georgia
  - Chiesi Clinical Trial - Site 840726, Stonecrest, Georgia
  - Chiesi Clinical Trial - Site 840564, Valdosta, Georgia
  - Chiesi Clinical Trial - Site 840724, Muncie, Indiana
  - Chiesi Clinical Trial - Site 840672, Zachary, Louisiana
  - Chiesi Clinical Trial - Site 840645, Annapolis, Maryland
  - Chiesi Clinical Trial - Site 840661, Baltimore, Maryland
  - Chiesi Clinical Trial - Site 840707, North Dartmouth, Massachusetts
  - Chiesi Clinical Trial - Site 840657, Troy, Michigan
  - Chiesi Clinical Trial - Site 840658, Port Gibson, Mississippi
  - Chiesi Clinical Trial - Site 840641, Saint Charles, Missouri
  - Chiesi Clinical Trial - Site 840714, St Louis, Missouri
  - Chiesi Clinical Trial - Site 840541, St Louis, Missouri
  - Chiesi Clinical Trial - Site 840669, St Louis, Missouri
  - Chiesi Clinical Trial - Site 840686, Omaha, Nebraska
  - Chiesi Clinical Trial - Site 840703, Henderson, Nevada
  - Chiesi Clinical Trial - Site 840529, Las Vegas, Nevada
  - Chiesi Clinical Trial - Site 840701, North Las Vegas, Nevada
  - Chiesi Clinical Trial - Site 840722, Bayonne, New Jersey
  - Chiesi Clinical Trial - Site 840667, Buffalo, New York
  - Chiesi Clinical Trial - Site 840678, New Windsor, New York
  - Chiesi Clinical Trial - Site 840520, New York, New York
  - Chiesi Clinical Trial - Site 840705, New York, New York
  - Chiesi Clinical Trial - Site 840626, The Bronx, New York
  - Chiesi Clinical Trial - Site 840604, The Bronx, New York
  - Chiesi Clinical Trial - Site 840664, Charlotte, North Carolina
  - Chiesi Clinical Trial - Site 840721, Charlotte, North Carolina
  - Chiesi Clinical Trial - Site 840610, Denver, North Carolina
  - Chiesi Clinical Trial - Site 840659, Gastonia, North Carolina
  - Chiesi Clinical Trial - Site 840540, Huntersville, North Carolina
  - Chiesi Clinical Trial - Site 840523, New Bern, North Carolina
  - Chiesi Clinical Trial - Site 840708, Shelby, North Carolina
  - Chiesi Clinical Trial - Site 840621, Winston-Salem, North Carolina
  - Chiesi Clinical Trial - Site 840627, Cincinnati, Ohio
  - Chiesi Clinical Trial - Site 840713, Columbus, Ohio
  - Chiesi Clinical Trial - Site 840647, Dayton, Ohio
  - Chiesi Clinical Trial - Site 840646, Toledo, Ohio
  - Chiesi Clinical Trial - Site 840668, Oklahoma City, Oklahoma
  - Chiesi Clinical Trial - Site 840692, Tulsa, Oklahoma
  - Chiesi Clinical Trial - Site 840671, Philadelphia, Pennsylvania
  - Chiesi Clinical Trial - Site 840683, Philadelphia, Pennsylvania
  - Chiesi Clinical Trial - Site 840578, Anderson, South Carolina
  - Chiesi Clinical Trial - Site 840592, Charleston, South Carolina
  - Chiesi Clinical Trial - Site 840528, Fort Mill, South Carolina
  - Chiesi Clinical Trial - Site 840598, North Charleston, South Carolina
  - Chiesi Clinical Trial - Site 840696, Rock Hill, South Carolina
  - Chiesi Clinical Trial - Site 840660, Franklin, Tennessee
  - Chiesi Clinical Trial - Site 840546, Franklin, Tennessee
  - Chiesi Clinical Trial - Site 840553, Knoxville, Tennessee
  - Chiesi Clinical Trial - Site 840535, Baytown, Texas
  - Chiesi Clinical Trial - Site 840634, Boerne, Texas
  - Chiesi Clinical Trial - Site 840704, Carrollton, Texas
  - Chiesi Clinical Trial - Site 840566, Cypress, Texas
  - Chiesi Clinical Trial - Site 840706, Dallas, Texas
  - Chiesi Clinical Trial - Site 840716, Houston, Texas
  - Chiesi Clinical Trial - Site 840698, Houston, Texas
  - Chiesi Clinical Trial - Site 840574, Kerrville, Texas
  - Chiesi Clinical Trial - Site 840551, McKinney, Texas
  - Chiesi Clinical Trial - Site 840575, Mesquite, Texas
  - Chiesi Clinical Trial - Site 840741, North Richland Hills, Texas
  - Chiesi Clinical Trial - Site 840663, Pearland, Texas
  - Chiesi Clinical Trial - Site 840609, Plano, Texas
  - Chiesi Clinical Trial - Site 840673, San Antonio, Texas
  - Chiesi Clinical Trial - Site 840681, San Antonio, Texas
  - Chiesi Clinical Trial - Site 840711, San Antonio, Texas
  - Chiesi Clinical Trial - Site 840729, San Antonio, Texas
  - Chiesi Clinical Trial - Site 840597, San Antonio, Texas
  - Chiesi Clinical Trial - Site 840600, Sherman, Texas
  - Chiesi Clinical Trial - Site 840552, Sugar Land, Texas
  - Chiesi Clinical Trial - Site 840526, Tomball, Texas
  - Chiesi Clinical Trial - Site 840693, Portsmouth, Virginia
  - Chiesi Clinical Trial - Site 840709, Everett, Washington
  - Chiesi Clinical Trial - Site 840562, Morgantown, West Virginia
  - Chiesi Clinical Trial - Site 840532, Greenfield, Wisconsin
- Argentina (24):
  - Chiesi Clinical Trial - Site 32502, Buenos Aires
  - Chiesi Clinical Trial - Site 32510, Buenos Aires
  - Chiesi Clinical Trial - Site 32515, Buenos Aires
  - Chiesi Clinical Trial - Site 32565, Buenos Aires
  - Chiesi Clinical Trial - Site 32514, Ciudad Autonoma Buenos Aires
  - Chiesi Clinical Trial - Site 32567, Ciudad Autonoma Buenos Aires
  - Chiesi Clinical Trial - Site 32507, Ciudad Autónoma de Buenos Aire
  - Chiesi Clinical Trial - Site 32563, Concepción del Uruguay
  - Chiesi Clinical Trial - Site 32503, Córdoba
  - Chiesi Clinical Trial - Site 32509, Córdoba
  - Chiesi Clinical Trial - Site 32501, Florida
  - Chiesi Clinical Trial - Site 32562, Mar del Plata
  - Chiesi Clinical Trial - Site 32505, Mendoza
  - Chiesi Clinical Trial - Site 32511, Mendoza
  - Chiesi Clinical Trial - Site 32513, Mendoza
  - Chiesi Clinical Trial - Site 32506, Quilmes
  - Chiesi Clinical Trial - Site 32553, Rosario
  - Chiesi Clinical Trial - Site 32508, San Juan Bautista
  - Chiesi Clinical Trial - Site 32512, San Miguel de Tucumán
  - Chiesi Clinical Trial - Site 32551, San Miguel de Tucumán
  - Chiesi Clinical Trial - Site 32561, San Miguel de Tucumán
  - Chiesi Clinical Trial - Site 32564, San Miguel de Tucumán
  - Chiesi Clinical Trial - Site 32566, San Rafael
  - Chiesi Clinical Trial - Site 32556, Santa Fe
- Austria (5):
  - Chiesi Clinical Trial - Site 40502, Feldbach
  - Chiesi Clinical Trial - Site 40504, Grieskirchen
  - Chiesi Clinical Trial - Site 40501, Linz
  - Chiesi Clinical Trial - Site 40503, Linz
  - Chiesi Clinical Trial - Site 40505, Wels
- Bosnia and Herzegovina (13):
  - Chiesi Clinical Trial - Site 70553, Banja Luka
  - Chiesi Clinical Trial - Site 70555, Bihać
  - Chiesi Clinical Trial - Site 70554, Bijeljina
  - Chiesi Clinical Trial - Site 70557, Foča
  - Chiesi Clinical Trial - Site 70556, Gradiška
  - Chiesi Clinical Trial - Site 70560, Mostar
  - Chiesi Clinical Trial - Site 70562, Mostar
  - Chiesi Clinical Trial - Site 70559, Sarajevo
  - Chiesi Clinical Trial - Site 70561, Sarajevo
  - Chiesi Clinical Trial - Site 70551, Travnik
  - Chiesi Clinical Trial - Site 70558, Trebinje
  - Chiesi Clinical Trial - Site 70563, Tuzla
  - Chiesi Clinical Trial - Site 70552, Zenica
- Bulgaria (25):
  - Chiesi Clinical Trial - Site 100535, Blagoevgrad
  - Chiesi Clinical Trial - Site 100534, Dimitrovgrad
  - Chiesi Clinical Trial - Site 100525, Gabrovo
  - Chiesi Clinical Trial - Site 100523, Haskovo
  - Chiesi Clinical Trial - Site 100533, Kozloduy
  - Chiesi Clinical Trial - Site 100527, Lovech
  - Chiesi Clinical Trial - Site 100515, Montana
  - Chiesi Clinical Trial - Site 100532, Pernik
  - Chiesi Clinical Trial - Site 100522, Pleven
  - Chiesi Clinical Trial - Site 100529, Plovdiv
  - Chiesi Clinical Trial - Site 100537, Razgrad
  - Chiesi Clinical Trial - Site 100512, Rousse
  - Chiesi Clinical Trial - Site 100516, Rousse
  - Chiesi Clinical Trial - Site 100536, Sevlievo
  - Chiesi Clinical Trial - Site 100501, Sofia
  - Chiesi Clinical Trial - Site 100509, Sofia
  - Chiesi Clinical Trial - Site 100514, Sofia
  - Chiesi Clinical Trial - Site 100517, Sofia
  - Chiesi Clinical Trial - Site 100518, Sofia
  - Chiesi Clinical Trial - Site 100530, Sofia
  - Chiesi Clinical Trial - Site 100531, Sofia
  - Chiesi Clinical Trial - Site 100538, Sofia
  - Chiesi Clinical Trial - Site 100524, Stara Zagora
  - Chiesi Clinical Trial - Site 100519, Vidin
  - Chiesi Clinical Trial - Site 100557, Vidin
- Chile (7):
  - Chiesi Clinical Trial - Site 152506, Concepción
  - Chiesi Clinical Trial - Site 152507, Quillota
  - Chiesi Clinical Trial - Site 152503, Santiago
  - Chiesi Clinical Trial - Site 152504, Santiago
  - Chiesi Clinical Trial - Site 152508, Santiago
  - Chiesi Clinical Trial - Site 152509, Talca
  - Chiesi Clinical Trial - Site 152501, Valparaíso
- Croatia (13):
  - Chiesi Clinical Trial - Site 191562, Dubrovnik
  - Chiesi Clinical Trial - Site 191552, Karlovac
  - Chiesi Clinical Trial - Site 191557, Osijek
  - Chiesi Clinical Trial - Site 191561, Rijeka
  - Chiesi Clinical Trial - Site 191563, Rijeka
  - Chiesi Clinical Trial - Site 191553, Sisak
  - Chiesi Clinical Trial - Site 191558, Split
  - Chiesi Clinical Trial - Site 191555, Zadar
  - Chiesi Clinical Trial - Site 191551, Zagreb
  - Chiesi Clinical Trial - Site 191554, Zagreb
  - Chiesi Clinical Trial - Site 191556, Zagreb
  - Chiesi Clinical Trial - Site 191559, Zagreb
  - Chiesi Clinical Trial - Site 191560, Zagreb
- Czechia (10):
  - Chiesi Clinical Trial - Site 203551, Brandýs nad Labem
  - Chiesi Clinical Trial - Site 203518, Havlíčkův Brod
  - Chiesi Clinical Trial - Site 203501, Jindřichův Hradec
  - Chiesi Clinical Trial - Site 203517, Měšice
  - Chiesi Clinical Trial - Site 203504, Miroslav
  - Chiesi Clinical Trial - Site 203516, Mladá Boleslav
  - Chiesi Clinical Trial - Site 203505, Prague
  - Chiesi Clinical Trial - Site 203507, Prague
  - Chiesi Clinical Trial - Site 203513, Prague
  - Chiesi Clinical Trial - Site 203515, Prague
- Estonia (3):
  - Chiesi Clinical Trial - Site 372553, Narva
  - Chiesi Clinical Trial - Site 372551, Tallinn
  - Chiesi Clinical Trial - Site 372552, Tartu
- Germany (21):
  - Chiesi Clinical Trial - Site 276505, Berlin
  - Chiesi Clinical Trial - Site 276506, Berlin
  - Chiesi Clinical Trial - Site 276510, Berlin
  - Chiesi Clinical Trial - Site 276511, Berlin
  - Chiesi Clinical Trial - Site 276515, Berlin
  - Chiesi Clinical Trial - Site 276556, Cottbus
  - Chiesi Clinical Trial - Site 276509, Darmstadt
  - Chiesi Clinical Trial - Site 276503, Delitzsch
  - Chiesi Clinical Trial - Site 276504, Frankfurt am Main
  - Chiesi Clinical Trial - Site 276557, Geesthacht
  - Chiesi Clinical Trial - Site 276501, Hamburg
  - Chiesi Clinical Trial - Site 276513, Hamburg
  - Chiesi Clinical Trial - Site 276514, Hamburg
  - Chiesi Clinical Trial - Site 276558, Hanover
  - Chiesi Clinical Trial - Site 276517, Koblenz
  - Chiesi Clinical Trial - Site 276502, Leipzig
  - Chiesi Clinical Trial - Site 276516, Leipzig
  - Chiesi Clinical Trial - Site 276551, Leipzig
  - Chiesi Clinical Trial - Site 276507, Mainz
  - Chiesi Clinical Trial - Site 276508, Munich
  - Chiesi Clinical Trial - Site 276518, Peine
- Greece (6):
  - Chiesi Clinical Trial - Site 300506, Athens
  - Chiesi Clinical Trial - Site 300504, Chortiatis
  - Chiesi Clinical Trial - Site 300501, Heraklion
  - Chiesi Clinical Trial - Site 300503, Ioannina
  - Chiesi Clinical Trial - Site 300505, Thessaloniki
  - Chiesi Clinical Trial - Site 300507, Volos
- Hungary (12):
  - Chiesi Clinical Trial - Site 348506, Balassagyarmat
  - Chiesi Clinical Trial - Site 348501, Budapest
  - Chiesi Clinical Trial - Site 348505, Csorna
  - Chiesi Clinical Trial - Site 348512, Edelény
  - Chiesi Clinical Trial - Site 348508, Gödöllő
  - Chiesi Clinical Trial - Site 348509, Monor
  - Chiesi Clinical Trial - Site 348507, Nyíregyháza
  - Chiesi Clinical Trial - Site 348513, Pécs
  - Chiesi Clinical Trial - Site 348552, Sellye
  - Chiesi Clinical Trial - Site 348510, Szeged
  - Chiesi Clinical Trial - Site 348503, Szombathely
  - Chiesi Clinical Trial - Site 348515, Törökbálint
- Israel (10):
  - Chiesi Clinical Trial - Site 376502, Ashkelon
  - Chiesi Clinical Trial - Site 376501, Beersheba
  - Chiesi Clinical Trial - Site 376511, Hadera
  - Chiesi Clinical Trial - Site 376508, Haifa
  - Chiesi Clinical Trial - Site 376510, Haifa
  - Chiesi Clinical Trial - Site 376503, Jerusalem
  - Chiesi Clinical Trial - Site 376506, Jerusalem
  - Chiesi Clinical Trial - Site 376507, Kfar Saba
  - Chiesi Clinical Trial - Site 376504, Ramat Gan
  - Chiesi Clinical Trial - Site 376509, Tel Aviv
- Latvia (8):
  - Chiesi Clinical Trial - Site 371557, Balvi
  - Chiesi Clinical Trial - Site 371553, Daugavpils
  - Chiesi Clinical Trial - Site 371554, Daugavpils
  - Chiesi Clinical Trial - Site 371555, Jūrmala
  - Chiesi Clinical Trial - Site 371558, Rēzekne
  - Chiesi Clinical Trial - Site 371551, Riga
  - Chiesi Clinical Trial - Site 371552, Riga
  - Chiesi Clinical Trial - Site 371556, Riga
- Mexico (10):
  - Chiesi Clinical Trial - Site 484502, Chihuahua City
  - Chiesi Clinical Trial - Site 484510, Chihuahua City
  - Chiesi Clinical Trial - Site 484505, Córdoba
  - Chiesi Clinical Trial - Site 484506, Cuauhtémoc
  - Chiesi Clinical Trial - Site 484501, Guadalajara
  - Chiesi Clinical Trial - Site 484507, Guadalajara
  - Chiesi Clinical Trial - Site 484509, Guadalajara
  - Chiesi Clinical Trial - Site 484503, Monterrey
  - Chiesi Clinical Trial - Site 484511, Monterrey
  - Chiesi Clinical Trial - Site 484504, Veracruz
- Netherlands (4):
  - Chiesi Clinical Trial - Site 528501, Beek
  - Chiesi Clinical Trial - Site 528504, Breda
  - Chiesi Clinical Trial - Site 528502, Heerlen
  - Chiesi Clinical Trial - Site 528505, Leeuwarden
- New Zealand (3):
  - Chiesi Clinical Trial - Site 554504, Christchurch
  - Chiesi Clinical Trial - Site 554502, Hamilton
  - Chiesi Clinical Trial - Site 554503, Tauranga
- North Macedonia (7):
  - Chiesi Clinical Trial - Site 807555, Bitola
  - Chiesi Clinical Trial - Site 807559, Gevgelija
  - Chiesi Clinical Trial - Site 807557, Ohrid
  - Chiesi Clinical Trial - Site 807553, Shtip
  - Chiesi Clinical Trial - Site 807552, Skopje
  - Chiesi Clinical Trial - Site 807554, Skopje
  - Chiesi Clinical Trial - Site 807556, Skopje
- Poland (15):
  - Chiesi Clinical Trial - Site 616518, Bialystok
  - Chiesi Clinical Trial - Site 616504, Giżycko
  - Chiesi Clinical Trial - Site 616515, Katowice
  - Chiesi Clinical Trial - Site 616522, Katowice
  - Chiesi Clinical Trial - Site 616509, Krakow
  - Chiesi Clinical Trial - Site 616511, Krakow
  - Chiesi Clinical Trial - Site 616514, Krakow
  - Chiesi Clinical Trial - Site 616503, Lodz
  - Chiesi Clinical Trial - Site 616523, Lodz
  - Chiesi Clinical Trial - Site 616519, Ostrowiec Świętokrzyski
  - Chiesi Clinical Trial - Site 616506, Poznan
  - Chiesi Clinical Trial - Site 616508, Poznan
  - Chiesi Clinical Trial - Site 616501, Sosnowiec
  - Chiesi Clinical Trial - Site 616502, Torun
  - Chiesi Clinical Trial - Site 616554, Wroclaw
- Romania (17):
  - Chiesi Clinical Trial - Site 642510, Bacau
  - Chiesi Clinical Trial - Site 642551, Brasov
  - Chiesi Clinical Trial - Site 642502, Cluj-Napoca
  - Chiesi Clinical Trial - Site 642504, Cluj-Napoca
  - Chiesi Clinical Trial - Site 642512, Cluj-Napoca
  - Chiesi Clinical Trial - Site 642554, Cluj-Napoca
  - Chiesi Clinical Trial - Site 642506, Cluj-Napoca Cluj
  - Chiesi Clinical Trial - Site 642508, Cluj-Napoca Cluj
  - Chiesi Clinical Trial - Site 642501, Constanța
  - Chiesi Clinical Trial - Site 642509, Craiova
  - Chiesi Clinical Trial - Site 642511, Craiova
  - Chiesi Clinical Trial - Site 642514, Iași
  - Chiesi Clinical Trial - Site 642503, Oradea
  - Chiesi Clinical Trial - Site 642513, Reșca
  - Chiesi Clinical Trial - Site 642505, Timișoara
  - Chiesi Clinical Trial - Site 642507, Timișoara
  - Chiesi Clinical Trial - Site 642515, Timișoara
- Russia (23):
  - Chiesi Clinical Trial - Site 643517, Kazan'
  - Chiesi Clinical Trial - Site 643513, Moscow
  - Chiesi Clinical Trial - Site 643528, Moscow
  - Chiesi Clinical Trial - Site 643516, Nizhny Novgorod
  - Chiesi Clinical Trial - Site 643503, Odintsovskiy
  - Chiesi Clinical Trial - Site 643504, Saint Petersburg
  - Chiesi Clinical Trial - Site 643505, Saint Petersburg
  - Chiesi Clinical Trial - Site 643506, Saint Petersburg
  - Chiesi Clinical Trial - Site 643508, Saint Petersburg
  - Chiesi Clinical Trial - Site 643510, Saint Petersburg
  - Chiesi Clinical Trial - Site 643511, Saint Petersburg
  - Chiesi Clinical Trial - Site 643512, Saint Petersburg
  - Chiesi Clinical Trial - Site 643514, Saint Petersburg
  - Chiesi Clinical Trial - Site 643519, Saint Petersburg
  - Chiesi Clinical Trial - Site 643520, Saint Petersburg
  - Chiesi Clinical Trial - Site 643531, Saint Petersburg
  - Chiesi Clinical Trial - Site 643515, Saratov
  - Chiesi Clinical Trial - Site 643525, Saratov
  - Chiesi Clinical Trial - Site 643521, Ulyanovsk
  - Chiesi Clinical Trial - Site 643502, Voronezh
  - Chiesi Clinical Trial - Site 643524, Vsevolozhsk
  - Chiesi Clinical Trial - Site 643507, Yaroslavl
  - Chiesi Clinical Trial - Site 643518, Yaroslavl
- Serbia (21):
  - Chiesi Clinical Trial - Site 688552, Belgrade
  - Chiesi Clinical Trial - Site 688553, Belgrade
  - Chiesi Clinical Trial - Site 688555, Belgrade
  - Chiesi Clinical Trial - Site 688557, Belgrade
  - Chiesi Clinical Trial - Site 688558, Belgrade
  - Chiesi Clinical Trial - Site 688559, Belgrade
  - Chiesi Clinical Trial - Site 688561, Belgrade
  - Chiesi Clinical Trial - Site 688569, Belgrade
  - Chiesi Clinical Trial - Site 688570, Jagodina
  - Chiesi Clinical Trial - Site 688564, Kamenitz
  - Chiesi Clinical Trial - Site 688566, Kamenitz
  - Chiesi Clinical Trial - Site 688556, Kragujevac
  - Chiesi Clinical Trial - Site 688562, Leskovac
  - Chiesi Clinical Trial - Site 688554, Niš
  - Chiesi Clinical Trial - Site 688568, Niš
  - Chiesi Clinical Trial - Site 688567, Pančevo
  - Chiesi Clinical Trial - Site 688560, Paraćin
  - Chiesi Clinical Trial - Site 688551, Sombor
  - Chiesi Clinical Trial - Site 688571, Sremska Mitrovica
  - Chiesi Clinical Trial - Site 688563, Užice
  - Chiesi Clinical Trial - Site 688565, Valjevo
- Slovakia (3):
  - Chiesi Clinical Trial - Site 703501, Bardejov
  - Chiesi Clinical Trial - Site 703503, Košice
  - Chiesi Clinical Trial - Site 703502, Spišská Nová Ves
- South Korea (11):
  - Chiesi Clinical Trial - Site 408556, Anyang-si
  - Chiesi Clinical Trial - Site 408551, Daegu
  - Chiesi Clinical Trial - Site 408560, Dongjak
  - Chiesi Clinical Trial - Site 408554, Gwangju
  - Chiesi Clinical Trial - Site 408559, Haeundae
  - Chiesi Clinical Trial - Site 408557, Incheon
  - Chiesi Clinical Trial - Site 408558, Incheon
  - Chiesi Clinical Trial - Site 408555, Jeonju
  - Chiesi Clinical Trial - Site 408552, Seoul
  - Chiesi Clinical Trial - Site 408553, Seoul
  - Chiesi Clinical Trial - Site 408561, Suwon,Gyeonggi-do
- Spain (6):
  - Chiesi Clinical Trial - Site 724503, Barcelona
  - Chiesi Clinical Trial - Site 724501, Córdoba
  - Chiesi Clinical Trial - Site 724505, Madrid
  - Chiesi Clinical Trial - Site 724551, Madrid
  - Chiesi Clinical Trial - Site 724504, Majadahonda
  - Chiesi Clinical Trial - Site 724502, Zaragoza
- Turkey (Türkiye) (9):
  - Chiesi Clinical Trial - Site 792512, Adana
  - Chiesi Clinical Trial - Site 792510, Bornova
  - Chiesi Clinical Trial - Site 792551, Çanakkale
  - Chiesi Clinical Trial - Site 792507, Istanbul
  - Chiesi Clinical Trial - Site 792514, Kocaeli
  - Chiesi Clinical Trial - Site 792513, Mersin
  - Chiesi Clinical Trial - Site 792506, Pamukkale
  - Chiesi Clinical Trial - Site 792508, Pendik
  - Chiesi Clinical Trial - Site 792511, Yenişehir
- Ukraine (20):
  - Chiesi Clinical Trial - Site 804522, Dnipro
  - Chiesi Clinical Trial - Site 804502, Ivano-Frankivsk
  - Chiesi Clinical Trial - Site 804504, Kharkiv
  - Chiesi Clinical Trial - Site 804505, Kharkiv
  - Chiesi Clinical Trial - Site 804506, Kharkiv
  - Chiesi Clinical Trial - Site 804509, Kharkiv
  - Chiesi Clinical Trial - Site 804503, Kherson
  - Chiesi Clinical Trial - Site 804511, Kiev
  - Chiesi Clinical Trial - Site 804520, Kremenchuk
  - Chiesi Clinical Trial - Site 804501, Kyiv
  - Chiesi Clinical Trial - Site 804508, Kyiv
  - Chiesi Clinical Trial - Site 804512, Kyiv
  - Chiesi Clinical Trial - Site 804516, Kyiv
  - Chiesi Clinical Trial - Site 804518, Kyiv
  - Chiesi Clinical Trial - Site 804521, Kyiv
  - Chiesi Clinical Trial - Site 804527, Odesa
  - Chiesi Clinical Trial - Site 804507, Poltava
  - Chiesi Clinical Trial - Site 804515, Vinnytsia
  - Chiesi Clinical Trial - Site 804517, Vinnytsia
  - Chiesi Clinical Trial - Site 804528, Zaporizhia
- United Kingdom (4):
  - Chiesi Clinical Trial - Site 826510, Belfast
  - Chiesi Clinical Trial - Site 826509, Bradford
  - Chiesi Clinical Trial - Site 826511, London
  - Chiesi Clinical Trial - Site 826512, Rochdale

IPD SHARING:
Plan to Share IPD: No